CLINICAL TRIAL: NCT02604576
Title: Efficacy of Fixed-dose Combination of Bromopride and Simethicone Versus Isolated Bromopride in Participants With Functional Dyspepsia.
Brief Title: Efficacy of Bromopride and Simethicone Versus Bromopride in Functional Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRDEMS1011
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Dyspepsia
Keywords: functional dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Simethicone; bromopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): FDC Bromopride 10 mg and Simethicone 80 mg
  Interventions: Drug: FDC Bromopride 10 mg and Simethicone 80 mg
- Group 2 (Active Comparator): Bromopride 10 mg (Digesan ® - Sanofi Aventis)
  Interventions: Drug: Bromopride 10 mg

INTERVENTIONS:
Drug: FDC Bromopride 10 mg and Simethicone 80 mg — Fixed-dose combination of Bromopride 10 mg and Simethicone 80 mg
  Other Names: Bromopride 10 mg and Simethicone 80 mg
  Arms: Group 1
Drug: Bromopride 10 mg — Bromopride 10 mg
  Other Names: Digesan®
  Arms: Group 2

SUMMARY:
Multi-center, randomized, superiority, double blind clinical trial to asses the efficacy of fixed-dose combination of bromopride and simethicone versus isolated bromopride on research participants diagnosed with functional dyspepsia.

DETAILED DESCRIPTION:
Multi-center, randomized, superiority, double blind clinical trial to asses the efficacy of fixed-dose combination of bromopride and simethicone versus isolated bromopride in the relief os dyspepsia symptoms on research participants diagnosed with functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent;
* Participants aged 18- 70 years;
* Clinical diagnosis of functional dyspepsia according to Rome III criteria;
* Minimum score of 22 points in PADYQ questionnaire

Exclusion Criteria:

* Diagnosis of gastroesophageal reflux disease, irritable bowel syndrome, inflammatory bowel disease, gallstones, strongyloidiasis, giardiasis or ascariasis, clinical disease or significant psychological;
* Positive diagnosis for Helicobacter pylori;
* Clinically significant organic diseases in the HDE (High Digestive Endoscopy) prior to randomization;
* History of esophageal surgery, gastrointestinal or other intra-abdominal surgery;
* Hypersensitivity to the components of the formulations;
* Allergy tartrazine yellow dye;
* Allergy to aspirin;
* Use of PPIs, H2 blockers, prokinetics, antibiotics, prostaglandins or bismuth salts in the last week before the screening visit;
* Use of NSAIDs or aspirin more than two days a week (except AAS <325mg / day), other drugs that induce gastrointestinal symptoms;
* Pregnant women or women without adequate contraception;
* Advance Participation in clinical trial protocols in the last twelve (12) months (CNS Resolution 251 of August 7, 1997, Part III, subsection J), unless the investigator considers that there may be direct benefit to it;
* Changes in hematological and biochemical tests: hemoglobin less than 12 g / dl, results with value 2 times the reference for AST, ALT, Gamma GT and alkaline phosphatase;
* Diagnosis of neurological or psychiatric diseases or decompensated diabetes;
* Use of drugs with anticholinergic action, narcotic analgesics, sedatives, hypnotics or tranquilizers;
* Alcoholism or sporadic use of alcohol and illicit drug use.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Symptoms assessed by proportion of participants who have reduction equal to or greater than 50% in symptoms through questionnaire PADYQ | 4 weeks

SECONDARY OUTCOMES:
Adverse events | 4 weeks
  Safety assessment will be performed by evaluating the incidence of adverse events in each group as well as the relationship of these events to the drug used, the amount and severity of reported events.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fernando Francesconi, MD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (10):
- Brazil (10):
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Centro de Medicina Reprodutiva Carlos Isaia Filho Ltda, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - AFIP, São Paulo, Sâo Paulo
  - UNIFAG, Bragança Paulista, São Paulo
  - Loema, Campinas, São Paulo
  - Instituto de Pesquisa Clinica de Campinas, Campinas, São Paulo
  - Allergisa, Campinas, São Paulo
  - Centro de Estudos Clínicos do Interior Paulista, Jaú, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo